CLINICAL TRIAL: NCT02305641
Title: Post-Marketing Surveillance of Kadcyla in Breast Cancer
Brief Title: An Observational Study of Kadcyla Safety in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29629
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Method of continuous surveillance per standard of care

SUMMARY:
This is a phase IV, prospective, multicenter, non-interventional study (regulatory post-marketing surveillance) in approximately 500 patients who are to receive Kadcyla (trastuzumab emtansine). Patients administered Kadcyla infusion at physician's discretion will be registered for this surveillance in Korea. Patients will be asked to provide informed consent; data will be collected by electronic Case Report Forms for approximately 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are administered with Kadcyla at physician's discretion will be registered for this study. The use of Kadcyla in the patients must fall into the approved indication in Korea.

Exclusion Criteria:

* Patients not receiving treatment for breast cancer with Kadcyla according to standard of care and in line with the current summary of product characteristics (SPC)/local labeling.
* A pediatric patient (age ≤18 years)
* Hypersensitivity for Kadcyla or any ingredient in this product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients administered Kadcyla infusion at physician's discretion
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Safety (composite outcome measure): Incidence of serious adverse events (SAEs), adverse drug reactions (ADRs); unexpected adverse events and ADRs; expected ADRs; non-serious ADRs | Up to 8 years

SECONDARY OUTCOMES:
Efficacy (composite outcome measure): Tumor response to Kadcyla treatment including complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- South Korea (38):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center; Surgical Department of Breast and Internal Secretion, Daegu
  - Chungnam National University Hospital, Daejeon
  - Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do
  - Bucheon St Mary's hospital, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Catholic Kwandong University International St. Mary'S Hospital., Incheon
  - Chonbuk National Uni Hospital, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Presbyterian Medical Center, Jeonju
  - Wonkwang University School of Medicine & Hospital, Jeonlabuk-do
  - NHIC Ilsan Hospital, Kyonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Korea Cancer Center Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hosiptal, Ulsan